CLINICAL TRIAL: NCT04118608
Title: Rhabdomyolysis - a Study of Patients and Laboratory Values to Guide Treatment
Acronym: RhabdoGuide
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other); Diakonhjemmet Hospital (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Mari Asphjell Bjørnaas, Project manager, Oslo University Hospital
Other Study IDs: 2019/370
Record Dates: First submitted 2019-09-20; First posted 2019-10-08 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Rhabdomyolysis is a potentially life-threatening syndrome characterized by breakdown of skeletal muscle, and leakage of intracellular substances such as myoglobin and creatine kinase (CK) into the circulation. The aetiological spectrum of rhabdomyolysis is extensive, and the clinical spectrum varies from a transient subclinical increase in CK activity to acute kidney injury (AKI) as a serious complication. There are no large prospective studies and only a few retrospective studies on rhabdomyolysis.

DETAILED DESCRIPTION:
Rhabdomyolysis is a potentially life-threatening syndrome characterized by breakdown of skeletal muscle, and leakage of intracellular substances such as myoglobin and creatine kinase (CK) into the circulation. The aetiological spectrum of rhabdomyolysis is extensive, and the clinical spectrum varies from a transient subclinical increase in CK activity to acute kidney injury (AKI) as a serious complication. There are no large prospective studies and only a few retrospective studies on rhabdomyolysis.

The project will give much needed information about incidence, aetiologies and the clinical course of rhabdomyolysis. The main objective will be to study rhabdomyolysis with focus on the development of AKI and how laboratory values can guide treatment, and thus act as basis for guidelines. More knowledge is needed about rhabdomyolysis and long-term kidney injury, and the study will aim to identify a risk population for later kidney injury, thus being able to refer this group to follow-up and prevent further injury. On the other hand, exercise-induced rhabdomyolysis patients are probably hospitalized more than necessary these days, and over-treatment could be prevented if better guidelines were obtained. The possible cardiotoxicity of myoglobin needs further study, and would benefit the patient group but also fill a knowledge gap for the clinicians. Therefore, this project will ideally obtain new knowledge for the health services, potentially improve existing practice and fill important knowledge gaps.

ELIGIBILITY:
1. Main study:

   * Inclusion Criteria: Patients age 18 years and older, with a muscle injury developed before hospitalization and serum CK activity ≥5000 U/L and/or serum myoglobin concentrations ≥1000 ng/ml within 72 hours after admission will be included.
   * Exclusion Criteria: Patients with unknown identity will be excluded.
2. Sub-study on rhabdomyolysis and cardiac enzymes:

   * Inclusion Criteria: All patients with troponins over 14 ng/L and who otherwise fulfills the inclusion criteria can be included.
   * Exclusion Criteria: Acute coronary syndrome, heart failure, arrythmia, previous myocarditis, circulatory shock, acute pulmonary embolism, thoracic trauma/heart trauma or CKD before hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective observational cohort study on patients with rhabdomyolysis admitted to emergency departments. Both medical and surgical/trauma departments will be included.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Development of Acute Kidney Injury (AKI) | Change of creatinine from baseline (KDIGO 2012 guidelines) through hospitalization (average 1 week)
  AKI will be defined according to KDIGO 2012 guidelines
Kidney function after three months and development of Chronic Kidney Disease (CKD) | 3 months
  Change in kreatinine and/or eGFR. CKD classifications followed KDIGO stages I-V

SECONDARY OUTCOMES:
Other complications | During hospitalization (average 1 week)
  Other complications including death
Risk stratification based on Myoglobin/Creatine kinase ratio | Change of creatinine from baseline (KDIGO 2012 guidelines) through hospitalization (average 1 week)
  Risk of AKI (see above) can be predicted based on this ratio
Association between rhabdomyolysis, elevated cardiac enzymes and the effect on myocardium. | Through hospitalization (average 1 week)
  Increased Troponin T levels and findings on echocardiography with strain and in some cardiac IMR
Risk stratification based on Myoglobin and Creatine kinase | Through hospitalization (average 1 week)
  See if risk of AKI (see above) can be predicted based on this

CONTACTS AND LOCATIONS:
Overall Officials: Vangstad, Principal Investigator — University of Oslo
Locations (1):
- Oslo University Hospital, Ullevaal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vangstad M, Gulsvik AK, Kro Birkeland JA, Ervik RL, Brekke FB, Akkouh OA, Jacobsen D, Bjornaas MA. Myoglobin-to-creatine kinase ratio enhances prediction of acute kidney injury in rhabdomyolysis. Emerg Med J. 2026 Jan 28:emermed-2025-215470. doi: 10.1136/emermed-2025-215470. Online ahead of print. PMID 41605622